CLINICAL TRIAL: NCT01737450
Title: A Phase II, Multicenter Trial Aiming to Evaluate the Clinical Interest of a Monotherapy With BKM120 , a Phosphoinositide 3-kinase (PI3K) Inhibitor in Patient With Metastatic Head and Neck Cancer Recurrent or Progressive Under Platin and Cetuximab-based Chemotherapy
Brief Title: Activity and Safety Study of BKM120 in Monotherapy in Patient With Metastatic Head and Neck Cancer Recurrent or Progressive
Acronym: PIK-ORL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government); Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET12-034; 2012-002403-18 (EudraCT Number)
Record Dates: First submitted 2012-11-13; First posted 2012-11-29 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Neoplasms; Neoplasm Metastasis; Recurrent Disease; Progressive Disease
Keywords: Metastatic head and neck cancer; PI3K inhibitor; Recurrent head and meck cancer; Progressive head and neck cancer; BKM120
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis; Recurrence; Disease Progression | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 (Experimental): Full dose=100 mg/day (oral route) One study cycle equals 28 days. Patients will be treated until disease progression, unacceptable toxicity, or willingness to stop.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120
  Other Names: Buparlisib

SUMMARY:
The aim of this study is to determine the activity, to assess the safety and tolerance of BKM120 in adult patients with recurrent or metastatic head and neck cancer progressive under platin and cetuximab-based chemotherapy.

DETAILED DESCRIPTION:
BKM120 is a PI3K inhibitor. The PI3K/Protein kinase B (AKT) signalling pathway deregulation is frequently observed in Head and neck cancer. In addition to its role in tumor genesis, the PI3K/AKT pathway seems to be involved in resistance to cetuximab.

In this context, the study proposal is to evaluate the clinical interest of a monotherapy with a PI3K inhibitor (BKM120, Novartis) in patients with metastatic head and neck cancers refractory or relapsing under platin and cetuximab based- chemotherapy. Since resistance to cetuximab can result from phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) mutation, PIK3CA amplification or mutation upstream in the PI3K pathway, BKM120 activity will be evaluated in two parallel independent cohorts of patients: patients presenting a PI3KCA mutation and patients without a PI3KCA mutation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult men and women ≥ 18 years at the day of inform consent signature.
* 2. Patients with metastatic or relapsed squamous cell head and neck carcinoma .
* 3. Documented progression or relapse after platin and cetuximab or anti-epidermal growth factor receptor (EGFR) -based chemotherapy at time of study drug start
* 4. Documented mutational status of PIK3CA before study drug start
* 5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 .
* 6. At least one measurable lesion by CT-scan as per RECIST 1.1 .
* 7. Life expectancy > 12 weeks.
* 8. Patients must be able to swallow capsules.
* 9. Adequate bone marrow, renal and liver function as defined by the following tests :
* Absolute neutrophil count ≥ 1.0 x 109/L,
* Platelet count > 100 x 109/L,
* Haemoglobin value above 9 g/dL,
* international normalized ratio (INR) ≤ 1.5
* Serum Creatinine ≤ 1.5 upper limit of normal (ULN)
* Glomerular filtration rate calculated using Cockcroft-Gault formula > 60ml/min (or MDRD formula for patients older than 65 years)
* Potassium, calcium, magnesium within normal limits for the institution
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < ULN (or < 3.0 x ULN if liver metastases are present))
* Serum bilirubin within normal range (or ≤ 1.5 ULN if liver metastases are present; or total bilirubin ≤ 3.0 ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
* Fasting plasma glucose (FPG) ≤ 120 mg/dL or ≤ 6.7 mmol/L.
* 10. Women of childbearing potential (entering the study after a confirmed menstrual period and who have a negative pregnancy test within ≤ 72 hours before initiating study treatment) must agree to use two methods of medically acceptable forms of contraception during the whole treatment period and for 1 month (= 5 x t½ of BKM120) after the last treatment intake.
* 11. Fertile males must use a highly effective contraception during dosing of any study agent + [5 x t1/2] + 12 weeks = contraception through 16 weeks after final dose of study therapy and should not father a child in this period. Female partner of male study subject: highly effective contraception during dosing of study agent + 4 weeks after final dose of study therapy
* 12. Patient should be able and willing to comply with study visits and procedures as per protocol.
* 13. Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.
* 14. Patients must be covered by a medical insurance.

Exclusion Criteria:

* 1. Patient having received previous treatment with PI3K and/or mammilian target of rapamycin (mTOR) inhibitors.
* 2. Patient with symptomatic central nervous system (CNS) metastases.
* 3. Patient with a concurrent malignancy or has a malignancy within 3 years of study enrollment, (with the exception of adequately treated basal or squamous cell carcinoma or non-melanomatous skin cancer).
* 4. Patient has any of the following mood disorders as judged by the Investigator or a Psychiatrist:
* Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others),
* Patients with active severe personality disorders (defined according to Diagnostic and Statistical Manual (DSM) - IV) are not eligible.

Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug.

* ≥ CTCAE grade 3 anxiety,
* or meets the cut-off score of ≥ 12 in the Patient Health Questionnaire (PHQ) -9 or a cut-off of ≥ 15 in the generalized anxiety disorder (GAD) -7 mood scale, respectively,
* or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9).
* 5. Patient concurrently using other approved or investigational anti-neoplasic agent.
* 6. Patient who has received anticancer therapy < 2 weeks or investigational treatment < 4 weeks prior the initiation of study drug.
* 7. Patient who has received radiotherapy ≤ 4 weeks prior to starting study drug or who have not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia).
* 8. Patient having had major surgery within 14 days prior to starting study drug or has not recovered from major side effects of the surgery.
* 9. Patient with poorly controlled diabetes mellitus (i.e. HbA1c > 8 %)
* 10. Patient with active cardiac disease including any of the following:
* Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO),
* corrected QT interval (QTc) > 480 (female) or 470 msec (male) on screening ECG (using the corrected QT Fridericia (QTcF) formulae),
* Angina pectoris that requires the use of anti-anginal medication,
* Ventricular arrhythmias except for benign premature ventricular contractions,
* Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication,
* Conduction abnormality requiring a pacemaker,
* Valvular disease with documented compromise in cardiac function,
* Symptomatic pericarditis.
* 11. Patient with a history of cardiac dysfunction including any of the following:
* Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function,
* History of documented congestive heart failure (New York Heart Association functional classification III-IV),
* Documented cardiomyopathy,
* Other cardiac arrhythmia not controlled with medication.
* 12. Patient currently receiving treatment with QT prolonging medication known to have a risk to induce Torsades de Pointes, and if the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* 13. Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120
* 14. Patient receiving chronic treatment (> 5 days) with steroids or another immunosuppressive agent. Note: Topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular) are allowed. Patients with previously treated brain metastases, who are on a stable low dose corticosteroids treatment (e.g., dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment, are eligible.
* 15. Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate her participation in the clinical study
* 16. Patient has a history of non-compliance to medical regimen.
* 17. Patient is currently being treated with drugs known to be strong inhibitors or inducers of isoenzyme Cytochrome P450 family 3 subfamily A member 4 (CYP3A), and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* 18. Patient has a known history of HIV infection.
* 19. Pregnant or nursing (lactating) woman.
* 20. Patient has a known hypersensitivity to any of the excipients of BKM120.
* 21. Patient has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy.
* 22. Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin, or fondaparinux is allowed.
* 23. Patient has acute viral hepatitis or a history of chronic or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, typically defined by elevated AST/ALT (persistent or intermittent), high HBV DNA level, HBsAg positive, or high HCV RNA level (testing not mandatory)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
2 months disease control rate | 2 months after the first BKM120 intake
  Control rate= Complete response, partial response and stable disease according to RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival | At 2 months, 4 months and then every 2 months
Overall survival (OS) | Baseline, at 2 months, 4 months and then every 2 months at the end of Study
  OS will be measured from the date of inclusion to the date of death from any cause.
Safety | continuous up to 30 days after the last treatment
  The assessment of safety will be based mainly on the frequency of adverse events based on the common toxicity criteria adverse event (CTCAE) V4.0 grade.
Objective response rate | At Baseline, 2 months, 4 months and then every 2 months, at the end of Study
  Objective response rate is defined as the proportion of patient with complete or partial response according RECIST 1.1
Duration of response | At Baseline, 2 months, 4months and then every 2 months, at the end of Study
  The duration of response will be measured from the time of first documented response until the first documented disease progression or death due to underlying cancer.
Time to Progression | At Baseline, 2 months, 4months and then every 2 months, at the end of Study
  Time to Progression will be measured from the time of treatment start until the first documented disease progression. Patients with no event at the time of the analysis will be censored at their last tumor assessment date.

CONTACTS AND LOCATIONS:
Overall Officials: Jérome FAYETTE, MD, Principal Investigator — Centre Léon Bérard, Lyon- FRANCE
Locations (9):
- France (9):
  - Hopital St André, Bordeaux
  - Hôpital BEAUJON, Clichy
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Centre Val d'Aurelle - Paul Lamarque, Montpellier
  - Centre Antoine LACASSAGNE, Nice
  - Institut Curie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Graupera M, Guillermet-Guibert J, Foukas LC, Phng LK, Cain RJ, Salpekar A, Pearce W, Meek S, Millan J, Cutillas PR, Smith AJ, Ridley AJ, Ruhrberg C, Gerhardt H, Vanhaesebroeck B. Angiogenesis selectively requires the p110alpha isoform of PI3K to control endothelial cell migration. Nature. 2008 May 29;453(7195):662-6. doi: 10.1038/nature06892. Epub 2008 Apr 30. PMID 18449193
- [Background] Schnell CR, Stauffer F, Allegrini PR, O'Reilly T, McSheehy PM, Dartois C, Stumm M, Cozens R, Littlewood-Evans A, Garcia-Echeverria C, Maira SM. Effects of the dual phosphatidylinositol 3-kinase/mammalian target of rapamycin inhibitor NVP-BEZ235 on the tumor vasculature: implications for clinical imaging. Cancer Res. 2008 Aug 15;68(16):6598-607. doi: 10.1158/0008-5472.CAN-08-1044. PMID 18701483
- [Background] Vokes EE, Weichselbaum RR, Lippman SM, Hong WK. Head and neck cancer. N Engl J Med. 1993 Jan 21;328(3):184-94. doi: 10.1056/NEJM199301213280306. No abstract available. PMID 8417385
- [Background] Saranath D, Panchal RG, Nair R, Mehta AR, Sanghavi VD, Deo MG. Amplification and overexpression of epidermal growth factor receptor gene in human oropharyngeal cancer. Eur J Cancer B Oral Oncol. 1992 Oct;28B(2):139-43. doi: 10.1016/0964-1955(92)90043-z. PMID 1306731
- [Background] Burtness B. The role of cetuximab in the treatment of squamous cell cancer of the head and neck. Expert Opin Biol Ther. 2005 Aug;5(8):1085-93. doi: 10.1517/14712598.5.8.1085. PMID 16050785